CLINICAL TRIAL: NCT03317067
Title: Effects of Dexmedetomidine on Delirium Duration of Non-intubated ICU Patients (4D Trial)
Acronym: 4D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU- 356; 2017-000731-14 (Other: 2017-000731-14)
Record Dates: First submitted 2017-10-09; First posted 2017-10-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Delirium; Agitation
Keywords: Dexmdetomidine; Haloperidol; Delirium; Productive Delirium; Agitation; Intubation; Ventilatory free days; Sedation; ICU patients; Mechanical Ventilation
MeSH Terms: conditions — Delirium; Psychomotor Agitation | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine (Experimental): Patients in the Dexmedetomidine (interventional) group will be treated with a continuous infusion of dexmedetomidine in case of agitated delirium.
  Interventions: Drug: Dexmedetomidine
- Normal Saline (NaCl 0.9%) (Placebo Comparator): Patients in the Normal Saline (control) group will be treated with a continuous infusion of normal saline in case of agitated delirium.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — The 4D trial is an investigator-initiated, prospective, multicenter, randomized, double-blinded, two-arm trial, randomizing 300 non-intubated ICU patients with diagnosis of agitated delirium to receive dexmedetomidine or placebo as a cure
  Arms: dexmedetomidine
Other: Placebo — The 4D trial is an investigator-initiated, prospective, multicenter, randomized, double-blinded, two-arm trial, randomizing 300 non-intubated ICU patients with diagnosis of agitated delirium to receive dexmedetomidine or placebo as a cure
  Arms: Normal Saline (NaCl 0.9%)

SUMMARY:
The primary purpose of the study is to evaluate whether dexmedetomidine is effective in treating agitated delirium of non-intubated ICI patients

DETAILED DESCRIPTION:
Delirium during intensive care unit (ICU) stay is frequent and associated with significant morbidity, mortality and healthcare related costs. International guidelines suggest its prevention. However, curative treatment remains unclearly established. Despite a non-unequivocal literature, haloperidol is the first line recommended neuroleptic. Dexmedetomidine, an alpha2-adrenergic receptors agonist has shown its efficiency in the treatment of delirium in intubated patients but also in its prevention. Dexmedetomidine represents a widely used alternative to haloperidol. Only few studies have compared the efficacy of dexmedetomidine in non-intubated ICU patients as a first line curative treatment of delirium. Main objective of 4D trial is to demonstrate that dexmedetomidine decreases delirium duration compared to placebo.

The 4D trial is an investigator-initiated, prospective, multicenter, randomized, double-blinded, two-arm trial, randomizing 300 non-intubated ICU patients with diagnosis of agitated delirium to receive dexmedetomidine or placebo as a cure. The primary outcome measure is a composite of duration of agitation or delirium or the use of intubation with deep sedation and mechanical ventilation. Secondary outcomes include mortalities at 7 and 28 days, ICU length of stay and occurrence of adverse effects. The sample size will allow the detection of a 50% decrease of agitation duration (120 minutes), of an absolute reduction of delirium duration (1 day) and of a 50% relative decrease of intubation and mechanical ventilation, with a type 1 error rate of 1.8 % (error risk inflation due to components of composite) and power of 90 %, assuming a 15 % incidence of intubation and mechanical ventilation requirements, an agitation duration of 240 minutes and a delirium duration of 3 days. One hundred and 10 patients by group will be needed. A intermediate analysis is scheduled and requires the inclusion of 150 patients in each group.

The 4D trial may provide important data on the safety of commonly used sedative dexmedetomidine and could have a significant impact on future treatment of non-intubated ICU patients presenting with agitated delirium.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 18 years

  * Patient hospitalized in an ICU
  * Presenting a productive delirium according to the following criteria:
  * acute onset (<2h) and fluctuating course during the same day
  * alteration of cognitive functions: disorganization of thought (delirium of persecution, inability to reason logically), abnormal perceptions (hallucinations), memory impairments, temporal disorientation, non- or misrecognitions, difficulties in naming objects or writing)
  * in whom a simple cropping and non-medicated therapeutics are not sufficient to allow symptoms' resolution for few hours
  * CAM-ICU positive AND a RASS > +1
  * Non-intubated or extubated (> 24h)
  * No contraindication of dexmedetomidine or haloperidol uses

Exclusion Criteria:

* • Age <18 years

  * Administration of dexmedetomidine and/or clonidine during the 72 hours before inclusion
  * Contraindication to the use of Dexmedetomidine, clonidine or haloperidol (history of allergy, Parkinson's disease, oro-pharyngeal dysfunction, arterial hypotension or bradycardia, QTc interval prolongation, and hepatic or renal dysfunction), as mentioned in the Summaries of Product Characteristics
  * Neuropsychiatric pathology judged by the investigator as a potential source of bias (in particular: active drug addiction, psychosis...)
  * Parturient or breast-feeding woman
  * Protected major (guardianship)
  * Patient's or relative's refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
duration of agitation (in hours), defined by a RASS ≥ +1 | at day 1
duration of delirium (in days), defined by a positive CAM-ICU | at day 1
delay (in hours) between inclusion and intubation requirement to control delirium with deep sedation and mechanical ventilation | at day 1
  requirement of intubation to control delirium with deep sedation and mechanical ventilation

SECONDARY OUTCOMES:
Length of ICU stay (in days) | at day 1
Number of ventilator free days | at day 30
Adverse effects such as the occurence of pneumonia (following the ATS definitions) and/or septicemia | at day 30
Duration of mechanical restraint prescribed and carried out | at day 30
Occurrence of tachycardia | at day 30
Occurrence of hypotension requiring any vasopressor administration | at day 30
All-cause mortality | at day 30
All-cause mortality | at day 7

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GODET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Godet T, Louis C, Rieu B, De Jong A, Couhault P, Pradel G, Tete H, Bourguignon N, Borao L, Jabaudon M, Futier E, Jaber S, Pereira B, Chanques G, Constantin JM; 4D study group. Dexmedetomidine for treatment of hyperactive delirium in non-intubated ICU patients: the 4D randomized clinical trial. Intensive Care Med. 2025 Dec;51(12):2305-2317. doi: 10.1007/s00134-025-08135-1. Epub 2025 Oct 29. PMID 41160116
- [Derived] Louis C, Godet T, Chanques G, Bourguignon N, Morand D, Pereira B, Constantin JM; AZUREA network. Effects of dexmedetomidine on delirium duration of non-intubated ICU patients (4D trial): study protocol for a randomized trial. Trials. 2018 Jun 4;19(1):307. doi: 10.1186/s13063-018-2656-x. PMID 29866205